CLINICAL TRIAL: NCT02324595
Title: Minimally Invasive Interval Debulking Surgery in Ovarian Neoplasm: a Feasibility Study
Acronym: MISSION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Fagotti, Anna, M.D. (Individual); Fanfani, Francesco, M.D. (Individual); Salvatore Gueli Alletti (Unknown)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Director, Dip per la Tutela della Salute della Donna e della Vita Nascente, del Bambino e dell'Adolescente, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10279/14
Record Dates: First submitted 2014-06-17; First posted 2014-12-24 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Stage IV Ovarian Carcinoma; Effects of Chemotherapy; Peritoneal Cavity Cancer
Keywords: Ovarian Cancer; Laparoscopy; Neoadjuvant Chemotherapy; Robotic; Interval Debulking Surgery
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laparoscopic Interval Debulking Surgery (Experimental): Patients affected by advanced epithelial ovarian cancer already submitted to neoadjuvant chemotherapy with evidence of complete/partial response
  Interventions: Procedure: Laparoscopic interval debulking surgery

INTERVENTIONS:
Procedure: Laparoscopic interval debulking surgery — Diagnostic laparoscopy with a careful exploration of peritoneal cavity: if available a 5 mm "flexible tip" videolaparoscope will be used to explore all peritoneal recesses.For eligible patients,will be placed 3 5mm trocar in standard position for pelvic surgery:cytoreduction will consist in total/radical hysterectomy,bilateral salpingo-oophorectomy,radical omentectomy.If needed pelvic/upper peritonectomy will be performed:in these cases additional trocar can be placed in right or left subcostal spaces. All surgical procedure requested will have be carried out by laparoscopy/robotic or by laparotomy,in case of increased surgical risk or technical impossibility:the case will be registered as laparotomic conversion.At the end of surgical procedures residual tumor will be registered
  Other Names: Laparoscopy

SUMMARY:
Phase II multicentric study

DETAILED DESCRIPTION:
The aim of this prospective Phase II multicentric study is to assess feasibility and early complications rate of "total laparoscopic/robotic" interval debulking surgery in patients with a clinical complete/partial response to neoadjuvant chemotherapy for advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years,
* Advanced ovarian cancer submitted to neoadjuvant chemotherapy,
* Clinical or serological complete/partial response (RECIST; GCIG),
* PS ≤ 2 (ECOG),
* Informed consent

Exclusion Criteria:

* Borderline and non-epithelial ovarian tumors,
* Stable/progressive disease,
* ASA 3-4,
* Severe cardiopulmonary disease,
* BMI > 40

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Operative complication rate | 30 days
  Intra- and post-operative complication rate of total laparoscopic/robotic interval debulking surgery

SECONDARY OUTCOMES:
Progression Free survival | one year
  time to recurrence
Overall Survival | One year
  time to last follow up/death

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, Prof, Principal Investigator — Catholic University of the Sacred Heart
Locations (2):
- Italy (2):
  - Catholic University of Sacred Heart Rome,, Rome, Rome
  - Policlinico Agostino Gemelli, Rome, Rome

REFERENCES:
- [Derived] Gueli Alletti S, Bottoni C, Fanfani F, Gallotta V, Chiantera V, Costantini B, Cosentino F, Ercoli A, Scambia G, Fagotti A. Minimally invasive interval debulking surgery in ovarian neoplasm (MISSION trial-NCT02324595): a feasibility study. Am J Obstet Gynecol. 2016 Apr;214(4):503.e1-503.e6. doi: 10.1016/j.ajog.2015.10.922. Epub 2015 Oct 31. PMID 26529370